CLINICAL TRIAL: NCT03889873
Title: Evaluating Change in Drinking Identity as a Mechanism for Reducing Hazardous Drinking - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kristen Lindgren, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STUDY00006542; 1R01AA024732-01 (NIH)
Record Dates: First submitted 2019-03-14; First posted 2019-03-26 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Drinking; Excess, Habit (Continual); Identity, Social
Keywords: Drinking identity; Hazardous drinking; Social networks; Self-efficacy; Alcohol craving; Cognitive control; Narrative writing
MeSH Terms: conditions — Habits; Social Identification

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a condition to receive one of eight writing prompt variants in a 2x2x2 study design. There is also a within subjects component as participants complete the same writing prompt 3 times (once per week over a 3-week period).
Who Masked: Investigator
Masking Description: The PI, the project coordinator, and experimenters will not know which participants have been assigned to each condition. Outcomes are assessed via computer/online survey. There is no human outcome assessor in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Drinking; No network; First-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as a low-risk drinker and describe this future self; the prompt does not instruct to write about social network (important people, friends, family); participant will write using first-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Drinking; Network; First-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as a low-risk drinker and describe this future self; the prompt instructions include writing about social network (important people, friends, family); participant will write using first-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Drinking; No network; Third-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as a low-risk drinker and describe this future self; the prompt does not instruct to write about social network (important people, friends, family); participant will write using third-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Drinking; Network; Third-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as a low-risk drinker and describe this future self; the prompt instructions include writing about social network (important people, friends, family); participant will write using third-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Smartphone; No network; First-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as someone who has reduced their smartphone usage and describe this future self; the prompt does not instruct to write about social network (important people, friends, family); participant will write using first-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Smartphone; Network; First-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as someone who has reduced their smartphone usage and describe this future self; the prompt instructions include writing about social network (important people, friends, family); participant will write using first-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Smartphone; No network; Third-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as someone who has reduced their smartphone usage and describe this future self; the prompt does not instruct to write about social network (important people, friends, family); participant will write using third-person pronouns.
  Interventions: Behavioral: Narrative Writing
- Smartphone; Network; Third-person (Experimental): In this narrative writing task, the participant is asked to imagine him/herself as someone who has reduced their smartphone usage and describe this future self; the prompt instructions include writing about social network (important people, friends, family); participant will write using third-person pronouns.
  Interventions: Behavioral: Narrative Writing

INTERVENTIONS:
Behavioral: Narrative Writing — An writing task in which participants are given a description of a possible future self (that varies 3 factors: topic; drinking vs. smartphone; perspective: 1st vs. 3rd-person; and social network: specifically asked to be included vs. not specifically asked to be included). Participants are asked to imagine that future self vividly and to write about the thoughts and feeling describe themselves and their experiences, the characteristics they hope or wish they will ideally possess, the characteristics that they would need to have and the roles they will take on or things they will be doing. Participants are given 20 minutes to think and write. They will write and think about the same future on each of three lab-sessions (which occur at 1-week intervals).

SUMMARY:
The purpose of the proposed research is to evaluate whether changes in drinking identity (DI; how much one associates one's self with drinking) can reduce hazardous drinking (HD; heavy alcohol use and negative alcohol-related consequences) among current college students. The study seeks to explore whether manipulating DI among participants will have changes in self-efficacy, craving, and HD. If such an effect can be found, DI may be a mechanism for HD behavior change and will allow researchers to develop and improve interventions aimed at HD behaviors in high-risk young adults.

DETAILED DESCRIPTION:
Experimentally manipulate DI to increase self-efficacy, decrease alcohol craving and reduce HD. We will recruit 328 student hazardous drinkers and use an expressive writing task to manipulate their DI, the salience of their social network, and their writing perspective. The last factor is included because writing in a self-distanced (3rd person) vs. self-immersed (1st person) perspective has been linked to greater cognitive control. We will evaluate the manipulation's immediate effects on DI, self-efficacy, and craving. Participants will also complete two weekly follow-up "booster" sessions. Longer-term effects on DI, self-efficacy, craving and HD will be evaluated at additional 2-week, 1-month, and 3-month follow-ups.

With the outbreak of the COVID-19 pandemic, new subject enrollment was paused between March and September 2020. In light of the continued COVID-19 pandemic, the study team made the decision to move the in-person, lab-based session (where participants completed the writing task) to online sessions as of October 2020. With the move to online sessions, we have discontinued the cue reactivity task and the accompanying craving assessment. Inclusion criteria have shifted slightly -- we now explicitly require participants to be currently living in Washington State (this criterion was implicit in our previous criteria and procedures) . The structure of the study otherwise remains the same.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be full-time UW students, fluent in the English language, and recent (past week) drinkers who self-report drinking hazardously (i.e., score an 8 or above on the Alcohol Use Disorder Identification Test, AUDIT). Participants must also own a smartphone.

Exclusion Criteria:

* None.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 329 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Changes in Implicit Drinking identity | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  drinking identity implicit association test (IAT)
Changes in Explicit Drinking identity | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Alcohol Self-concept Scale; item responses range from -3 to +3; average score on all items is calculated; lower scores represent a better outcome
changes in self-efficacy | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  drinking refusal self-efficacy questionnaire
cue-related craving | Cue related craving will be assessed following the cue reactivity task, which occurs during the third and final lab-based session (technically, the third week of the study)
  current craving from cue reactivity task; assessed via alcohol urge questionnaire
changes in past week craving | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Penn Alcohol Craving Scale; item responses range from 0 to 6; total score on all items is calculated (can range from 0 to 30); lower scores = better outcome
changes in alcohol consumption | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Modified timeline follow back will assess past daily alcohol consumption (# standard drinks per day); higher consumption = worse outcomes
changes in last 3 month alcohol problems | Assessed at lab 1 (week1) and 3-month follow up; data will be reported through study completion (3 month follow up)
  Rutgers Alcohol Problems Inventory (RAPI) will be used to assess alcohol problems; item response options range from 0 to 4; total score ranges from 0 to 100; higher scores = worse outcomes
changes in last two week alcohol problems | assessed at lab 2 and 3 (weeks 2 and 3) and at 2 week and 1 month follow up; data will be reported through 1 month follow up
  adapted from RAPI & Young Adult Alcohol Problems Screening Test (YAAPST); item responses are 0 (did not happen) or 1 (happened); higher scores (range from 0 to 10) = worse outcomes

SECONDARY OUTCOMES:
changes in future drinking intentions | assessed at lab 1, lab 2, lab 3 (weeks 1-3); data will be reported through week 3
  adapted from daily drinking questionnaire; assesses how much individuals think they will drink each day of the next week
changes in frequency of heavy & extreme binge drinking | assessed at lab 1 (week 1) &
  frequency of heavy episodic (4/5 or more drinks for women/men on a single occasion) and extreme binge drinking (at least 8/10 drinks or at least 12/15 drinks for women/men on a single occasion); definitions are from the National Institute of Alcohol and Alcoholism
Changes in Readiness to Change Drinking | post-writing (lab 1, lab 2, lab 3) long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  single item about readiness to change one's drinking (from Rollnick, Mason, & Butler, 1999); ranges from 0 to 6; higher scores = more readiness to change one's drinking; higher scores = better outcome
Changes in single-item assessing self-efficacy to limit one's drinking | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Item developed by Cervone & Shadel; item ranges from 0 to10; higher scores = greater self-efficacy to limit one's drinking; higher scores = better outcome

OTHER OUTCOMES:
Changes in social network composition | will be assessed at baseline and 3-month follow up; data will be reported through study completion (3 month follow up)
  Important people measure will ask about the 10 most important individuals in one's social network, including whether or not each one drinks; the variables that are derived include the density of drinkers in the network; higher density = more drinkers (worse outcome)
Changes in desire thinking about alcohol | assessed at lab 1 (week 1) and long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Assessed via the Desire Thinking Questionnaire; response options range from 1 to 4; total scores (range from 10 to 40) indicate amount of desire thinking about alcohol; higher scores = more desire thinking (worse outcome)
Changes in smartphone addiction proneness | Assessed at lab 1 (week 1) and long-term follow up (2 week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Assessed via the smartphone addiction proneness scale; will use total score (sum); response options range from 1 to 4; total scores (range from 15 to 60), higher scores = more addiction proneness (worse outcome)
Changes in smartphone use | Assessed at lab 1 (week 1) and long-term follow up (2 week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  item assessing frequency of use and length of time not using; higher frequency of use = worse outcome; higher length of time not using = better outcome
changes in affect | assessed pre-post-writing during lab 1, lab 2, lab 3 (weeks 1-3); data will be reported through week 3
  State (current) affect will be assessed immediately prior to and after the narrative writing task; two items (one assessing positive affect and one assessing negative affect); item response range from 0 to 100, with 100 indicating greater intensity of feeling; affect will be assess each time participants complete the narrative writing task (i.e. lab 1, lab 2, lab 3); no changes in affect are expected
Manipulation check questions about the narrative writing task | will be assessed and reported for each of the 3 lab sessions (weeks 1, 2, and 3)
  Following the narrative writing task (which occurs at each of the lab session), participants will be asked 5 items about what they wrote and imagined; each item will be evaluated separately; response options range from -3 to +3; items assess how vividly they imagined what they wrote; how easy it was to imagine what they wrote; how much writing made them seem their life differently; how plausible what they imagined was; how relatable what they wrote about was; for all items higher scores = better outcomes
Changes in single-item assessing self-efficacy to limit one's smartphone use | will be assessed at lab 1, lab 2, lab 2 (weeks 1-3) & long-term follow up (2-week, 1 month, 3 month); data will be reported through study completion (3 month follow up)
  Item developed by Cervone & Shadel; item response options range from 0 to 10; higher scores = greater self-efficacy to limit one's smartphone use; higher scores = better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kristen P Lindgren, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share responses to questionnaires and writing exercises with co-investigators. We do not currently have plans to store data in a repository/database (for example, via the Open Science Framework [OSF] - https://osf.io/), though we may ultimately do so should this be a condition of publishing in a scientific journal or necessary for other unforeseen reasons. Should we do so, we would not publish or make available or the narrative writing responses verbatim. Similarly, we would also not publish or make available the variables that describe the 10 most important people on the important people measure. No direct identifiers will be included in any data shared.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available after the grant period of award is completed unless there is a requirement to make data publicly available as a condition of publication.
Access Criteria: Data access requests will be reviewed by the PI and study research coordinator. Requestors will be required to sign a data use agreement.